CLINICAL TRIAL: NCT01271517
Title: Effects of New Longacting Insulin Analogs on Metabolic Control, Endogenous Insulin Production, GH/IGF-I Axis and Quality of Life - Comparison of NPH, Glargine Och Detemir Insulin From the Debut of Type 1 Diabetes Mellitus in Adolescents
Brief Title: Basal Analog Study - Comparison of Lantus or Levemir With NPH Insulin From T1DM Diagnosis
Acronym: BAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Peter Bang, MD, PhD, Associated Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eudract-number 2005-001726-80
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Basal insulin; long acting insulin analogs; metabolic control; HbA1c; C-peptide; IGF-I; GH; IGFBP
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin, Isophane; Insulin Glargine; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulatard (Active Comparator): Treatment twice daily with Insulatard plus Novorapid at meals. Doses adjusted according to bloodsugars
  Interventions: Drug: NPH insulin
- Lantus (Active Comparator): Treatment once daily with Levemir plus Novorapid at meals. Doses adjusted according to bloodsugars
  Interventions: Drug: Glargine
- Levemir (Active Comparator): Treatment twice daily with Levemir plus Novorapid at meals. Doses adjusted according to bloodsugars
  Interventions: Drug: Detemir

INTERVENTIONS:
Drug: NPH insulin — Treatment twice daily with Insulatard plus Novorapid at meals. Doses adjusted according to bloodsugar
  Arms: Insulatard
Drug: Glargine — Treatment once daily with Lantus plus Novorapid at meals. Doses adjusted according to bloodsugars
  Arms: Lantus
Drug: Detemir — Treatment twice daily with Levemir plus Novorapid at meals. Doses adjusted according to bloodsugars
  Arms: Levemir

SUMMARY:
Hypothesis: Basal insulin analogs with continuous 24-hour delivery of insulin improve glycemic control during the first year of treatment of children/adolescents with type 1 diabetes mellitus (T1DM)by preserving endogenous insulin production and a close to normal balance of the GH-IGF-axis.

This a randomized, open-label, parallel-group trial of 120 children, 7 - 17 years of age, newly diagnosed with T1DM. The investigators will investigate whether the use of long-acting basal insulin analogs Lantus (Glargine) or Levemir (Detemir) during the first year of treatment results in improved glycemic control (HbA1c) compared with Insulatard (NPH insulin) when given in a meal insulin therapy regimen with rapid acting Novorapid (insulin aspart). The investigators will explore possible mechanisms of action by determining remaining endogenous insulin production and changes in the GH-IGF-axis. The investigators will also assess changes in body composition and evaluate quality of life in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes and novel to insulin therapy
* Age 7 - 17 years
* Informed consent

Exclusion Criteria:

* Moderate to severe ketoacidosis (pH<7.2 and/or standard bicarbonate <10 mmol/l)
* Suspected non-type 1
* IA2 and GAD65: all-antibody negative
* Celiac disease or other chronic disease
* Hypothyroidism, if not well controlled
* Syndromes
* Previous anorexia nervosa
* Neuro-psychiatric disease
* Malignancy

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2005-09; Primary Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 1 year
  The study compare HbA1c one year after start of treatment at diagnosis of T1DM in patients treated with Lantus or Levemir with patients treated with Insulatard.

SECONDARY OUTCOMES:
Stimulated C-peptide | 2 weeks and 3, 6 and 12 month
  Sustacal stimulated C-peptide after an overnight fast
IGF-I | diagnosis, 2 weeks, 3,6,9 and 12 month
  Serum IGF-I concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Pediatrics, Karolinska University Hospital, Stockholm, Sweden